CLINICAL TRIAL: NCT06092008
Title: Establishing and Implementing Pneumonia Diagnosis in ED Older Adults: A Mixed Methods Approach
Brief Title: Performance of New Diagnostic Methods in Older Adults With Pneumonia
Acronym: PNEUMO
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Katherine Buck, Assistant Professor, Ohio State University
Other Study IDs: 2022H0136
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Create a clinical diagnostic pathway for older ED adults with pneumonia and its subgroups (bacterial, viral, and co-infection) and determine whether novel biomarkers improve diagnostic accuracy. The investigators will conduct a prospective observational trial of 250 ED patients ≥65 years old with suspected pneumonia. The investigators will perform analyses overall and by subgroups, seeking common models to ease adoption.

ELIGIBILITY:
Inclusion Criteria:

- Adults aged 65 and older presenting to the ED with suspected pneumonia defined as (1) either a physician order for CXR OR CT OR a chief complaint consistent with dyspnea; AND (2) physician suspicion of pneumonia prior to ED testing (score of 2-5 on Likert scale)

Exclusion Criteria:

* inability to obtain consent from the patient or an LAR
* active cancer
* organ transplant
* immunosuppression
* trauma activation
* suicidal ideation
* incarceration
* antibiotics in the last 14 days
* a separate episode of lower respiratory illness in the last 30 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged 65 and older presenting to the Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Pneumonia | 3 years
  Presence or absence of pneumonia based on adjudicator review of chart. The goal of the study is to create a diagnostic pathway for pneumonia in older adult emergency department patients.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States